CLINICAL TRIAL: NCT05016076
Title: The Multi-Strategy Intervention to Enhance Quality of Anesthesia Care for Obese Patients: A Factorial Randomized Controlled Trial
Brief Title: Multi-Strategy Intervention for Anesthesia Care of Obese Patients A Factorial Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID outbreak in the community
Sponsor: YingHsuanTai (Other)
Responsible Party: Sponsor-Investigator, YingHsuanTai, Principal Investigator, Taipei Medical University Shuang Ho Hospital
Organization: Taipei Medical University Shuang Ho Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: JIRB-N202101039
Record Dates: First submitted 2021-08-07; First posted 2021-08-23 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Obesity; Bariatric Surgery Candidate; Tracheal Intubation Morbidity; Nausea and Vomiting, Postoperative; Hyperglycemia Drug Induced; Gastric Reflux
MeSH Terms: conditions — Obesity; Postoperative Nausea and Vomiting; Gastroesophageal Reflux | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dexamethasone (Active Comparator): In the designated patients, 8 mg of dexamethasone or placebo will be given intravenously within 10 minutes after the induction of anesthesia. Anesthesia will be maintained with 2-3 vol% sevoflurane and 60% oxygen in nitrogen, whereas the fraction of inspired oxygen (FiO2) 0.8-1.0 will be used during pneumoperitoneum to ensure oxygen saturation higher than 92%.
  Interventions: Drug: Dexamethasone 8 mg
- Placebo (0.9% sodium chloride) (Placebo Comparator): In the designated patients, 8 mg of dexamethasone or placebo will be given intravenously within 10 minutes after the induction of anesthesia. Anesthesia will be maintained with 2-3 vol% sevoflurane and 60% oxygen in nitrogen, whereas the fraction of inspired oxygen (FiO2) 0.8-1.0 will be used during pneumoperitoneum to ensure oxygen saturation higher than 92%.
  Interventions: Drug: Placebo (0.9% sodium chloride)
- Inspiratory pressure (10 cmH2O) (Active Comparator): After the loss of eyelash reflex, a Guedel oropharyngeal airway (Biçakcilar, Istanbul, Turkey) will be placed into the oral cavity to assure adequate mouth opening. A facemask will be applied firmly to the patient's face to ensure an adequate seal. A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea is determined by end-tidal capnography occurs, mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure, at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator.
  Interventions: Diagnostic Test: Applied inspiratory pressure (10, 15, 20, or 25 cmH2O)
- Inspiratory pressure (15 cmH2O) (Active Comparator): After the loss of eyelash reflex, a Guedel oropharyngeal airway (Biçakcilar, Istanbul, Turkey) will be placed into the oral cavity to assure adequate mouth opening. A facemask will be applied firmly to the patient's face to ensure an adequate seal. A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea is determined by end-tidal capnography occurs, mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure, at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator.
  Interventions: Diagnostic Test: Applied inspiratory pressure (10, 15, 20, or 25 cmH2O)
- Inspiratory pressure (20 cmH2O) (Active Comparator): After the loss of eyelash reflex, a Guedel oropharyngeal airway (Biçakcilar, Istanbul, Turkey) will be placed into the oral cavity to assure adequate mouth opening. A facemask will be applied firmly to the patient's face to ensure an adequate seal. A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea is determined by end-tidal capnography occurs, mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure, at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator.
  Interventions: Diagnostic Test: Applied inspiratory pressure (10, 15, 20, or 25 cmH2O)
- Inspiratory pressure (25 cmH2O) (Active Comparator): After the loss of eyelash reflex, a Guedel oropharyngeal airway (Biçakcilar, Istanbul, Turkey) will be placed into the oral cavity to assure adequate mouth opening. A facemask will be applied firmly to the patient's face to ensure an adequate seal. A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea is determined by end-tidal capnography occurs, mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure, at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator.
  Interventions: Diagnostic Test: Applied inspiratory pressure (10, 15, 20, or 25 cmH2O)
- Video intubating stylet (Active Comparator): A tracheal tube (ConvaTec, Berkshire, England, UK) in appropriate sizes is preloaded over the Trachway® video intubating stylet (TVI-4050, Markstein Sichtec Medical Corp, Taichung, Taiwan), which is introduced into oral cavity to visualize the epiglottis and guided to glottis via a monitor after full neuromuscular blockade is achieved.
  Interventions: Device: Tracheal intubation using video intubating stylet, video laryngoscopy, or direct laryngoscopy
- Video laryngoscopy (Active Comparator): A tracheal tube is preloaded over a GlideRite® stylet, which is specifically designed to work with GlideScope® video laryngoscope (Verathon Medical, Bothell, WA, USA). GlideScope® blade size 3 (GS-3) or 4 (GS-4) is used in all patients.
  Interventions: Device: Tracheal intubation using video intubating stylet, video laryngoscopy, or direct laryngoscopy
- Direct laryngoscopy (Active Comparator): Tracheal tubes are prepared with a hockey stick-shaped stylet, and direct laryngoscopy is performed using a size-3 or -4 Macintosh blade (Rüsch Inc., Duluth, GA, USA).
  Interventions: Device: Tracheal intubation using video intubating stylet, video laryngoscopy, or direct laryngoscopy
- Goal-directed hemodynamic therapy (Active Comparator): Subjects of the GDHT group will be managed according to the ERAS algorithm utilizing ProAQT® parameters to maintain the cardiac index ≥ 2.5 l·min-1·m-2.61 In brief, if cardiac index < 2.5 l·min-1·m-2, a bolus of 150 ml of crystalloid fluid will be given until the stroke volume variation is < 10%. If cardiac index < 2.5 l·min-1·m-2 despite the stroke volume variation of ≥ 10% following fluid challenge, continuous intravenous infusion of dopamine 5-10 μg·kg-1·min-1 will be administered. If mean arterial pressure is < 70 mmHg despite cardiac index ≥ 2.5 l·min-1·m-2, intravenous infusion of norepinephrine 2-10 μg·min-1 will be used.
  Interventions: Device: Goal-directed hemodynamic therapy targeting cardiac index
- Usual care (control) (No Intervention): Subjects allocated to the control group are hemodynamically managed as per anesthesiologist preference. Typically, isolated hypotension (20% decrease in mean arterial pressure below baseline or < 60 mmHg) is treated by single or consecutive boluses of norepinephrine 5 or 10 μg. If hypotension persists, repeat boluses of ephedrine 4 mg will be administered until mean arterial pressure is above 60 mmHg. If hypotension is accompanied by signs of hypovolemia (urine output < 0.5 ml·kg-1·hr-1 and/or an increase in heart rate > 20% above baseline), crystalloid or colloid fluids will be given until urine output and/or heart rate are normalized. If hypotension persists despite volume challenge, norepinephrine will be used.

INTERVENTIONS:
Drug: Dexamethasone 8 mg — In the designated patients, 8 mg of dexamethasone or placebo will be given intravenously within 10 minutes after the induction of anesthesia.
  Arms: Dexamethasone
Diagnostic Test: Applied inspiratory pressure (10, 15, 20, or 25 cmH2O) — A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea determined by end-tidal capnography occurs, a mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure (PEEP), at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator (Carestation 620, Datex-Ohmeda, Inc., Madison, WI, USA).
  Arms: Inspiratory pressure (10 cmH2O); Inspiratory pressure (15 cmH2O); Inspiratory pressure (20 cmH2O); Inspiratory pressure (25 cmH2O)
Device: Tracheal intubation using video intubating stylet, video laryngoscopy, or direct laryngoscopy — In video intubating stylet group, a tracheal tube (ConvaTec, Berkshire, England, UK) in appropriate sizes is preloaded over the Trachway® video intubating stylet (TVI-4050, Markstein Sichtec Medical Corp, Taichung, Taiwan), which is introduced into oral cavity to visualize the epiglottis and guided to glottis via a monitor after full neuromuscular blockade is achieved. In video laryngoscopy group, a tracheal tube is preloaded over a GlideRite® stylet, which is specifically designed to work with GlideScope® video laryngoscope (Verathon Medical, Bothell, WA, USA). GlideScope® blade size 3 (GS-3) or 4 (GS-4) is used in all patients. In direct laryngoscopy group, tracheal tubes are prepared with a hockey stick-shaped stylet, and direct laryngoscopy is performed using a size-3 or -4 Macintosh blade (Rüsch Inc., Duluth, GA, USA).
  Arms: Direct laryngoscopy; Video intubating stylet; Video laryngoscopy
Device: Goal-directed hemodynamic therapy targeting cardiac index — Subjects of the GDHT group will be managed according to the ERAS algorithm utilizing ProAQT® parameters to maintain the cardiac index ≥ 2.5 l·min-1·m-2. In brief, if cardiac index < 2.5 l·min-1·m-2, a bolus of 150 ml of crystalloid fluid will be given until the stroke volume variation is < 10%. If cardiac index < 2.5 l·min-1·m-2 despite the stroke volume variation of ≥ 10% following fluid challenge, continuous intravenous infusion of dopamine 5-10 μg·kg-1·min-1 will be administered. If mean arterial pressure is < 70 mmHg despite cardiac index ≥ 2.5 l·min-1·m-2, intravenous infusion of norepinephrine 2-10 μg·min-1 will be used.
  Arms: Goal-directed hemodynamic therapy
Drug: Placebo (0.9% sodium chloride) — Placebo of 0.9% sodium chloride will be given intravenously within 10 minutes after the induction of anesthesia.
  Arms: Placebo (0.9% sodium chloride)

SUMMARY:
The main objective of this study is to investigate the optimal anesthesia for obese patients undergoing bariatric surgery in the strategies of positive pulmonary ventilation, tracheal intubation technique, hemodynamic monitoring, and postoperative nausea and vomiting (PONV) prophylaxis, as the followed:

1. To evaluate the effectiveness and adverse effect of intravenous dexamethasone for PONV prophylaxis
2. To determine the safe inspiratory pressure to prevent the occurrence of gastric insufflation during facemask ventilation using point-of-care ultrasonography of antrum
3. To compare the effectiveness and safety between video intubating stylet and video laryngoscope in the placement of tracheal tubes
4. To apply minimally invasive CO monitors in guiding goal-directed hemodynamic therapy and assess its impact on major complications and postoperative recovery

DETAILED DESCRIPTION:
Substudy 1: An evaluation of the effect of intravenous dexamethasone on postoperative nausea and vomiting

At the operating room, participants will be initially placed in a ramped position and then moved into a reverse Trendelenburg position to achieve a 30-degree incline of the thorax before preoxygenation. Each participant will be randomly assigned 1:1, stratified by presence of diabetes mellitus, to one of each of the following two interventions: dexamethasone (8 mg intravenously) and placebo (0.9% sodium chloride). The envelopes of group allocation will be opened just before the induction of general anesthesia.

After preoxygenation using facemask with pure oxygen 10 l·min-1 until end-tidal fractional oxygen concentration in the expired air (EtO2) ≥ 80%, general anesthesia will be induced with propofol 1.5-2.0 mg·kg-1 ideal body weight and fentanyl 1-2 μg·kg-1 total body weight. Tracheal intubation will be facilitated with rocuronium 0.8-1.0 mg·kg-1 ideal body weight. After induction, a radial artery catheterization will be performed for continuous monitoring of arterial pressure and measurement of serum glucose. In the designated patients, 8 mg of dexamethasone or placebo will be given intravenously within 10 minutes after the induction of anesthesia. Anesthesia will be maintained with 2-3 vol% sevoflurane and 60% oxygen in nitrogen, whereas the fraction of inspired oxygen (FiO2) 0.8-1.0 will be used during pneumoperitoneum to ensure oxygen saturation higher than 92%. If the value of surgical pleth index (CARESCAPE B650 Monitor, GE Healthcare, Chicago, IL, USA) is more than 50 or heart rate or blood pressure increases by more than 20% from baseline values during surgery, an intravenous bolus of fentanyl 25 or 50 μg will be given. Besides, the concentration of sevoflurane can be adjusted as clinically appropriate.

After surgery, all participants will receive supplemental oxygen, and pain will be relieved with ketorolac 15 to 30 mg. The need for postoperative opioids will be at the discretion of the anesthesiologist, and the dose will be adjusted according to clinical needs. Participants who request rescue antiemetic therapy or who have an emetic episode will be given droperidol 1.25 mg. If symptoms persist, metoclopramide 10 mg will be administered.

Primary outcome is the incidence of PONV, which includes any nausea, emetic episodes (retching or vomiting), or both during the first 24 postoperative hour. At the 2nd and 24th postoperative hours, trained investigators who are blinded to the group allocation will record the number of emetic episodes, the time each one occurs, and self-reported worst nausea episode during the preceding duration on an 11-point scale (0: no nausea and 10: the most severe nausea).

Substudy 2: An investigation of the threshold inspiratory pressure for gastric insufflation using ultrasonography of gastric antrum

The investigators will measure the antral area of each participant lying in supine position on the operating table, using a portable ultrasound device (LOGIQ™, GE Healthcare, Chicago, IL, USA, fitted with a 1.5 to 5.0 MHz convex transducer). The investigators will determine the longitudinal (D1) and anteroposterior (D2) diameters of the cross-section of antrum in the sagittal plane passing through abdominal aorta.50 To obtain a standardized scanning level, the aorta and left lobe of the liver are employed as internal landmarks. The relaxed diameters of the antrum are measured between antral contractions. The area of gastric antrum is calculated using the formula: antral area = D1×D2×π / 4. In addition, the gastric fluid volume will be calculated with a validated model based on the cross-sectional area of the gastric antrum, described previously.51 Participants will be randomized into one of the four groups defined by the applied inspiratory pressure (10, 15, 20, or 25 cmH2O) using blocked randomization. During induction of anesthesia, normal saline 20 ml will be immediately infused after the administration of rocuronium 0.8-1.0 mg·kg-1 ideal body weight.52 After loss of eyelash reflex, a Guedel oropharyngeal airway (Biçakcilar, Istanbul, Turkey) will be placed into the oral cavity to assure adequate mouth opening. A facemask will be applied firmly to the patient's face to ensure an adequate seal. A two-handed head-tilt jaw-thrust maneuver will be performed to establish an open airway. Once apnea determined by end-tidal capnography occurs, a mechanical ventilation with the assigned peak inspiratory pressure will be initiated. The pressure-controlled mode will be used with an inspiratory-to-expiratory ratio of 1:2 and no positive end-expiratory pressure (PEEP), at a frequency of 15 breath·min-1 and with 100% oxygen, by the ventilator (Carestation 620, Datex-Ohmeda, Inc., Madison, WI, USA).53 Real-time ultrasonography of the antrum will be performed by the same anesthesiologist who performs the preoperative ultrasonography. Another anesthetist will perform continuous auscultation over epigastric area. The investigators performing ultrasonography and auscultation are blinded one to another regarding the detection of gastric insufflation and the inspiratory pressure of pressure-controlled ventilation. The ultrasonography screen will be concealed from the anesthetist performing the auscultation. Facemask ventilation will be continued for 2 min. The trachea will be thereafter intubated, and the antral area will be measured again.

Primary outcome is the episode of gastric insufflation. The ultrasonographic diagnosis of gastric insufflation is defined as the presence of an acoustic shadow phenomenon and/or a comet-tail artifact into the antrum.14 A typical whoosh sound with gurgling while auscultating over the epigastrium defines the diagnosis of gastric insufflation by auscultation method.54

Substudy 3: A comparison of video intubation stylet and video laryngoscope in tracheal intubation

Eligible participants will be randomly allocated 1:1:1, stratified by body mass index > 50 kg·m-2, to group 1 (video intubating stylet), group 2 (video laryngoscopy), or group 3 (direct laryngoscopy). Tracheal intubation will be performed by experienced attending anesthesiologists who have performed at least 100 cases each with Trachway® video intubating stylet, GlideScope® video laryngoscopy, and Macintosh direct laryngoscopy. The anesthesiologist performing tracheal intubation is blinded to all preoperative evaluations.

In group 1, a tracheal tube (ConvaTec, Berkshire, England, UK) in appropriate sizes is preloaded over the Trachway® video intubating stylet (TVI-4050, Markstein Sichtec Medical Corp, Taichung, Taiwan), which is introduced into oral cavity to visualize the epiglottis and guided to glottis via a monitor after full neuromuscular blockade is achieved. In group 2, a tracheal tube is preloaded over a GlideRite® stylet, which is specifically designed to work with GlideScope® video laryngoscope (Verathon Medical, Bothell, WA, USA). GlideScope® blade size 3 (GS-3) or 4 (GS-4) is used in all participants. In group 3, tracheal tubes are prepared with a hockey stick-shaped stylet, and direct laryngoscopy is performed using a size-3 or -4 Macintosh blade (Rüsch Inc., Duluth, GA, USA). In all participants, backward, upward, and rightward pressure on the larynx and Sellick maneuvers are allowable to obtain the best glottic view.55,56 If the initial intubation attempt fails or is terminated for desaturation (defined as SpO2 < 92%) or need to change the patient's position, the intubation device will be removed, and manual bag mask ventilation will be performed. Intubation failure is defined as more than three intubation attempts or need to change intubation devices. Any intubation rescue techniques will be used at the discretion of the staff anesthesiologist.

Primary outcome is the best glottis visualization, graded according to Cormack and Lehane's classification with external laryngeal pressure applied.57 Glottic views graded as III or IV are regarded as difficult.

Substudy 4: An investigation of the putative benefits of goal-directed hemodynamic therapy targeting cardiac index in obese patients undergoing laparoscopic sleeve gastrectomy

At the operation room, the investigators will apply the Masimo Radical 7 pulse oximetry (Masimo Corp., Irvine, CA, USA) to the fingers of all enrolled patients to measure perfusion index and SpO2 throughout the surgery. After the placement of a tracheal tube, patients will receive ventilator support with the tidal volume 6-8 ml·kg-1 ideal body weight, a respiratory rate of 10-15 min-1 and PEEP 5 cmH2O applied by the ventilator.60 The FiO2 will be set at 0.3-0.7 to maintain SpO2 ≥ 98% throughout the surgery. Each patient will be randomly allocated to one of each of the following two groups: goal-directed hemodynamic therapy and control.

In both groups, intraoperative maintenance rate of crystalloid fluids is 3 ml·kg-1·hr-1 ideal body weight. ProAQT®-derived hemodynamic data and peripheral perfusion index and SpO2 will be acquired at the following time points: 5 min after induction of anesthesia, 5 min after start of pneumoperitoneum and head-up tilting, 5 min after end of pneumoperitoneum, cessation of volatile anesthetics, and 5 min after extubation. Subjects of the GDHT group will be managed according to the ERAS algorithm utilizing ProAQT® parameters to maintain the cardiac index ≥ 2.5 l·min-1·m-2.61 In brief, if cardiac index < 2.5 l·min-1·m-2, a bolus of 150 ml of crystalloid fluid will be given until the stroke volume variation is < 10%. If cardiac index < 2.5 l·min-1·m-2 despite the stroke volume variation of ≥ 10% following fluid challenge, continuous intravenous infusion of dopamine 5-10 μg·kg-1·min-1 will be administered. If mean arterial pressure is < 70 mmHg despite cardiac index ≥ 2.5 l·min-1·m-2, intravenous infusion of norepinephrine 2-10 μg·min-1 will be used.

Subjects allocated to the control group are hemodynamically managed as per anesthesiologist preference. Typically, isolated hypotension (20% decrease in mean arterial pressure below baseline or < 60 mmHg) is treated by single or consecutive boluses of norepinephrine 5 or 10 μg. If hypotension persists, repeat boluses of ephedrine 4 mg will be administered until mean arterial pressure is above 60 mmHg. If hypotension is accompanied by signs of hypovolemia (urine output < 0.5 ml·kg-1·hr-1 and/or an increase in heart rate > 20% above baseline), crystalloid or colloid fluids will be given until urine output and/or heart rate are normalized. If hypotension persists despite volume challenge, norepinephrine will be used.

In both groups, the fluid, inotrope, and vasopressor responsiveness, ProAQT® parameters (cardiac index, stroke volume variation, systemic vascular resistance, and mean arterial pressure), and the signals of pulse oximetry (perfusion index and SpO2) will be evaluated and recorded for each 15-min interval throughout the surgery. In control group, the ProAQT® monitoring will be concealed from the anesthetist in charge. Artifact-free signals are considered valid for statistical analysis. At the end of surgery, all participants will receive a manual recruitment maneuver of 30 to 40 cmH2O for 10 s three times. In all patients, cessation of volatile anesthetics will be timed to facilitate early awakening after wound closure. All patients will be decurarized from rocuronium-induced neuromuscular blockade with sugammadex dosed at 2 mg·kg-1 ideal body weight + 40%.62 Primary outcome is a composite of major complications according to the European Perioperative Clinical Outcome definitions within 30 days after surgery, including myocardial ischemia or infarction, arrhythmia, acute kidney injury, gastrointestinal bleeding, anastomotic breakdown, surgical site infection, and hospital-acquired pneumonia.63

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years
2. Body mass index ≥ 30 kg·m-2
3. Undergoing laparoscopic sleeve gastrectomy at Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

Exclusion Criteria:

1. Pregnant or lactating women
2. Severe cardiopulmonary distress, including left ventricular ejection fraction < 40%, double or triple vessel disease, New York Heart Association functional classification ≥ 3, peripheral oxygen saturation by pulse oximetry (SpO2) < 90% in room air, and moderate to severe pulmonary hypertension.
3. Previous esophageal, gastric, or duodenal surgery.
4. Previous head and neck surgery or radiation therapy
5. Previous cervical spine injury
6. High-degree cardiac arrythmia, including atrial fibrillation and severe atrioventricular block
7. Use of cardiac pacemaker or automated implantable cardioverter defibrillator
8. Chronic kidney disease, stage ≥ 4 (estimated glomerular filtration rate < 30 ml·min-1)
9. Planned transferal to intensive care unit for mechanical ventilation
10. QTc prolongation determined by a standard 12-lead electrocardiogram
11. Patients using emetogenic or antiemetic drugs within 24 hours before surgery
12. Patients requiring rapid sequence induction or fiberoptic awake intubation
13. Patient refusal to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Substudy 1: Number of participants developing postoperative nausea and vomiting | The first 24 postoperative hour
  Primary outcome is postoperative nausea and vomiting, which includes any nausea, emetic episodes (retching or vomiting), or both during the first 24 postoperative hour. At the 2nd and 24th postoperative hours, trained investigators who are blinded to the group allocation will record the number of emetic episodes, the time each one occurs, and self-reported worst nausea episode during the preceding duration on an 11-point scale (0: no nausea and 10: the most severe nausea).
Substudy 2: The threshold inspiratory pressure for gastric insufflation | Within 2 min after induction of anesthesia
  Primary outcome is the episode of gastric insufflation. The ultrasonographic diagnosis of gastric insufflation is defined as the presence of an acoustic shadow phenomenon and/or a comet-tail artifact into the antrum. A typical whoosh sound with gurgling while auscultating over the epigastrium defines the diagnosis of gastric insufflation by auscultation method.
Substudy 3: The best glottis visualization, graded according to Cormack and Lehane's classification | From the induction of anesthesia to the 24th postoperative hours
  Primary outcome is the best glottis visualization, graded according to Cormack and Lehane's classification with external laryngeal pressure applied. The minimum and maximum values of Cormack and Lehane's grade are I and IV, respectively. Glottic views graded as III or IV are regarded as difficult.
Substudy 4: Number of participants developing postoperative major complications | Within 30 days after surgery
  Primary outcome is a composite of major complications according to the European Perioperative Clinical Outcome definitions within 30 days after surgery, including myocardial ischemia or infarction, arrhythmia, acute kidney injury, gastrointestinal bleeding, anastomotic breakdown, surgical site infection, and hospital-acquired pneumonia. Any events of the above complications will be determined and analyzed aggregately and separately.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Hsuan Tai, M.D., Principal Investigator — Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT05016076/Prot_SAP_000.pdf